CLINICAL TRIAL: NCT03403816
Title: Objective Assessment of Physical Activity in Before-school Physical Activity Programs
Acronym: BOKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Reebok Foundation (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angie Cradock, Senior Research Scientist, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-1224
Record Dates: First submitted 2017-12-20; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Physical Activity; Sleep
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Students in grades K-6 at 7 schools in two communities participating in a before school physical activity program offered at no cost to participating families that focuses on engaging elementary and middle school students in physical activity, skill development and brief nutrition education sessions.
  .
  Interventions: Behavioral: Before School Physical Activity Program
- Comparison (No Intervention): Students in grades K-6 at the same 7 schools in two communities as the intervention participants, but who did not participate in the before school physical activity program.

INTERVENTIONS:
Behavioral: Before School Physical Activity Program — BOKS is a before school physical activity program offered at no cost to participating families that focuses on engaging elementary and middle school students in physical activity, skill development and brief nutrition education sessions that prepare them for a day of learning. The BOKS curriculum includes 12 weeks of instruction and 40 minutes of structured kid-friendly activities that include warm-ups, skill of the week, running, relay and obstacle course activities and nutritional tips. The BOKS team provides training for BOKS leaders free of charge each month. BOKS is currently being used in more than 1,800 schools in the US and Canada.
  Other Names: Build Our Kids Success (BOKS)
  Arms: Intervention

SUMMARY:
This study will determine the effectiveness of a free before-school physical activity program, BOKS (Build Our Kids' Success), in increasing objectively measured physical activity levels among children in elementary and middle school in 7 schools in Massachusetts.

DETAILED DESCRIPTION:
This study will determine the effectiveness of a free before-school physical activity program, BOKS (Build Our Kids' Success), in increasing objectively measured physical activity levels among children in elementary and middle school in 7 schools in Massachusetts. The study focuses on capturing valid and objective assessments of student-level physical activity during BOKS program time and assessing the impact of the BOKS program on overall daily physical activity levels using minute-by-minute physical activity level data among elementary aged students. Data is also collected to understand how increasing physical activity may impact students' sleep.

ELIGIBILITY:
Inclusion Criteria:

* Attending public elementary and middle school in two selected Massachusetts communities with BOKS programming

Exclusion Criteria:

* None

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 432 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Total steps per day | Participants wore a Fitbit activity monitor for up to 5 school days beginning with the before school period simultaneously for 24 hours/day
  The primary outcome measure is a physical activity measure of how many steps per day participants took.

SECONDARY OUTCOMES:
Active minutes | Participants wore a Fitbit activity monitor for up to 5 school days beginning with the before school period simultaneously for 24 hours/day
  A secondary outcome measure is a measure of how many minutes participants spent in light, moderate and vigorous activity per day.
Sleep duration | Participants wore Fitbit activity monitors for 24 hours for up to 5 school days
  A secondary outcome measure is the amount of time participants spent asleep each night, measured by a Fitbit activity monitor, which collects a measure of total sleep time.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cradock AL, Barrett JL, Taveras EM, Peabody S, Flax CN, Giles CM, Gortmaker SL. Effects of a before-school program on student physical activity levels. Prev Med Rep. 2019 Jul 3;15:100940. doi: 10.1016/j.pmedr.2019.100940. eCollection 2019 Sep. PMID 31367511